CLINICAL TRIAL: NCT05922748
Title: Brain Injury and Cognitive Function: Neuropsychology and Neuroimaging
Brief Title: Brain Injury and Cognitive Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C13-41; 2013-A01207-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-06-14; First posted 2023-06-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Lesion; Cognitive Deficit Following Brain Lesions
Keywords: neuroimaging; cognitive deficit; MEG; EEG; MRI
MeSH Terms: conditions — Cognition Disorders | interventions — X-Rays; Evoked Potentials

STUDY DESIGN:
Intervention Model Description: We will study patients (n= 300) suffering from focal brain lesions and healthy control subjects (n= 600 for imaging, n= 600 for purely behavioural studies)
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patient (Experimental): suffering from brain damage
  Interventions: Other: imaging; Other: Evoked Potentials; Other: MEG; Behavioral: Behavioural tests
- healthy control subjects for imaging (Active Comparator): healthy control subjects for imaging
  Interventions: Other: imaging; Other: Evoked Potentials; Other: MEG; Behavioral: Behavioural tests
- healthy control subjects for purely behavioural studies (Active Comparator): healthy control subjects for purely behavioural studies
  Interventions: Other: imaging; Other: Evoked Potentials; Other: MEG; Behavioral: Behavioural tests

INTERVENTIONS:
Other: imaging — Brain activation is demonstrated by measuring signal changes in brain regions. Activations will be determined by comparison between conditions and in relation to periods of rest
  Other Names: MRI
Other: Evoked Potentials — EEG signals, referenced to the right mastoid, were digitised at 125 Hz with an elliptical low-pass input filter at 49 Hz
Other: MEG — MEG signals reflect changes in magnetic field evoked by changes in neuronal activity
Behavioral: Behavioural tests — Behavioural tests will be evaluated.

SUMMARY:
The objective of this exploratory study is to elucidate the underlying cerebral mechanisms of cognitive deficits. To achieve this, the investigator will apply functional brain imaging techniques to patients suffering from cognitive deficits due to cerebral lesions.

The investigator will employ a "single-case" approach, suitable for studying rare behavioral profiles such as acquired reading disorders (alexia) or visual perception impairments (agnosia). If necessary, the investigator will use multiple non-invasive imaging methods in the same patients, including:

1. Magnetic Resonance Imaging (structural and functional), renowned for its spatial resolution and the diverse information it provides, and
2. Electrophysiological methods (MEG and EEG), notable for their temporal resolution.

The employed stimuli will consist of visual or auditory presentations of verbal material (words, sentences, numbers, etc.), potentially combined with the collection of simple vocal or motor responses (button presses).

The results will be interpreted by integrating the neuropsychological analysis of the deficit and the lesion topography.

Importantly, following the methodology of single-case neuropsychology, the stimulation protocols will be modulated and adapted to each individual case. Consequently, parallel data should be collected from healthy control subjects whenever necessary.

For protocol development, the investigator will also collect purely behavioral data, without brain imaging, from groups of control subjects.

DETAILED DESCRIPTION:
The study of the cerebral mechanisms underlying mental functions, specifically in humans, relies on two sources of data: the study of patients with brain lesions and neuroimaging. While neuroimaging has experienced spectacular developments in recent years, allowing for the characterization of the functional properties of multiple brain systems, only the study of patients can establish the causal involvement of these regions in the processes at hand by observing the selective deficits resulting from lesions. This logic applies not only to acquired focal lesions resulting from, for example, vascular accidents or surgical resections but also to selective developmental cognitive disorders such as dyslexia or dyscalculia, which have been shown to result from focal abnormalities in brain development.

Over the years, research teams employing this protocol have successfully utilized both approaches, and in an innovative manner, combined them in studies exploring cognitive deficits using neuroimaging. For example, Gaillard et al. (2006) and Epelbaum et al. (2008) investigated reading disorders related to small cortical lesions by combining behavioral studies, anatomical MRI, diffusion tensor imaging (DTI) of white matter tracts, functional MRI, and intracerebral recordings of evoked potentials (EPs) in the same patient. The rarity of behavioral profiles such as acquired reading disorders motivates the use of an approach known as "single-case studies." Significant advancements in neuropsychology have only been made possible through the study of single cases. In such studies, one or a few patients are examined in great detail on an individual basis, and their behavior is compared to explicit cognitive models of the specific function under investigation. Consequently, alongside standardized test batteries, evaluation protocols must necessarily be tailored and adapted to each individual case. On the other hand, group studies are not feasible for rare behavioral profiles such as acquired reading disorders (alexia) or visual perception impairments (agnosia). This unique case approach can be greatly enhanced by brain imaging. This is now achievable due to the sufficient power of functional magnetic resonance imaging (fMRI), enabling the analysis of activations in a single subject. Similarly, advancements in recording and data processing techniques in evoked potentials (EP) and magnetoencephalography (MEG) allow the analysis of individual patient performances. Furthermore, the flexible adaptation of stimulation protocols to each patient necessitates parallel data collection from a few control subjects whenever required.

Therefore, the aim of this exploratory project is to continue this work in cognitive neuroimaging, with the specific objective of comparing the results obtained from multiple non-invasive imaging methods (fMRI, EEG, and MEG) applied to patients with cerebral lesions (and to control groups of subjects as needed). In fact, within the scope of our exploratory study, the investigator aim to investigate the spatiotemporal dynamics of brain activity involved in specific higher cognitive functions in humans: language comprehension and production, mental calculation, as well as conscious and unconscious perception. The investigator will individually assess patients selected based on the nature of their deficit and the topography of their lesions, along with control subjects. Neurological patients will be followed for one year after consenting, with multiple testing and neuroimaging sessions. Patients may withdraw from the study at any time. Control subjects should be comparable to the patients in terms of age and sociocultural level and will, therefore, be matched for these variables in each patient's case. They will receive auditory stimuli through headphones or visual stimuli presented on a screen and will perform elementary tasks (memorization, comprehension, classification, production, etc.), indicating the correct response verbally or using response buttons when necessary. The investigator may refer the same subjects to different types of examinations (MRI, EP, MEG) to compare their results, which will be interpreted by integrating the neuropsychological analysis of the deficit and lesion topography. The investigator reserve the option to employ only one or two of these imaging methods in certain subjects. Additionally a group of healthy volunteers will be tested, with only the collection of their behavioral responses.

ELIGIBILITY:
INCLUSION CRITERIA

Common criteria for patients and healthy volunteers:

* Age: 18 years and older
* Affiliation with a social security system
* Signed informed consent
* No psychotropic medication intake in the week prior to the examination, and no alcohol consumption on the eve of the examination (subjects will be instructed to have a good night's sleep before the examination).

Specific criteria for patients:

- Patients must present either cerebral lesions (vascular, malformative, tumoral) or traumatic injuries, or a history of neonatal or congenital conditions that may result in selective cognitive impairments, or congenital or acquired visual perception disorders.

NON INCLUSION CRITERIA

Common criteria for patients and volunteers:

* Pregnant, lactating, or postpartum women (except for purely behavioral tests).
* Individuals with visual or auditory deficits that would interfere with the tasks to be performed during brain imaging acquisition.
* Contraindications for MRI (except for purely behavioral tests):
* Cardiac or neural stimulation devices
* Ferromagnetic surgical clips
* Cochlear implants
* Intra-ocular metallic foreign bodies or objects in the nervous system
* Implants or metallic objects that may concentrate the radiofrequency field
* Lack of informed consent
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2014-02-05 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
MRI (Functional Magnetic Resonance Imaging) | 13 years
  Brain activation is revealed by measuring signal changes in brain regions. Activations will be determined by comparing conditions and compared to resting periods using analysis techniques.
MEG (Magnetoencephalography) | 13 years
  MEG signals reflect changes in the magnetic field evoked by neuronal activity. They are collected and analyzed using specific analysis methods.
ERPs (Event-Related Potentials) | 13 years
  EEG signals, referenced to the right mastoid, are digitized at 125 Hz with a low-pass elliptical input filter at 49 Hz.

CONTACTS AND LOCATIONS:
Locations (1):
- ICM - Paris Brain Institute, Paris, Île-de-France Region, France